CLINICAL TRIAL: NCT07365501
Title: Acute Effect of Nurse-assessed Remote Ischemic Preconditioning on Improving Vascular Parameters in Patients With Suspected Heart Failure With Preserved Ejection Fraction
Acronym: PIRIC-FEp
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Universidad Pontificia Comillas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ND
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HF - Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic preconditioning (Experimental): Participants randomized to the PIR intervention group will receive a hand-held blood pressure device (Welch Allyn DuraShock™ DS45, NY, USA) to self-administer PIR. The cuff will be placed around the upper arm and inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, and this cycle will be repeated another three times.
  Interventions: Procedure: remote ischemic preconditioning
- No remote ischemic preconditioning (No Intervention): No intervention

INTERVENTIONS:
Procedure: remote ischemic preconditioning — Participants randomized to the PIR intervention group will receive a hand-held blood pressure device (Welch Allyn DuraShock™ DS45, NY, USA) to self-administer PIR. The cuff will be placed around the upper arm and inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, and this cycle will be repeated another three times. The arm on which participants will apply the PIR is the left arm. Participants will be supervised during the PIR session by a nurse to ensure that it is performed correctly.
  Arms: remote ischemic preconditioning

SUMMARY:
The PIRIC-FEp study will be a randomized clinical trial in sedentary patients with suspected heart failure with preserved ejection fraction.

Objectives: 1) To evaluate the acute efficacy of remote ischemic preconditioning performed by nurses, a noninvasive cardioprotective intervention that uses cycles of ischemia and reperfusion in the extremities, in improving vascular parameters.

Methodology: Patients will be recruited in Health Centers in the city. Those assigned to the intervention group will wear a self-administered blood pressure cuff, inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, in repeated cycles four times. The control group will receive no intervention. All participants will be examined, at baseline, 0 minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention. Different vascular parameters will be evaluated, including peripheral and central Systolic and Blood Pressure, peripheral and central Mean Arterial Pressure, peripheral and central Pulse Pressure, Heart Rate, Cardiac Output, Stroke Volume, Peripheral Vascular Resistance, aortic Pulse Wave Velocity and Augmentation Index normalized to a heart rate of 75 beats per minute. The study will be approved by an Ethics Committee, participants will be informed and will have to sign a written consent. The statistical analysis will include three phases: verification of randomization, use of covariance models for dependent variables, and sensitivity analysis with propensity score matching. All analyses will be performed on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of HF (Clinical suspicion of HF)
2. Sedentary men and women (structured exercise <2 x 30 min/week).
3. Age ≥40 years
4. Written informed consent
5. Clinically stable for 6 weeks
6. Optimal medical treatment for ≥6 weeks.

Exclusion Criteria:

1. Non-cardiac causes of HF symptoms:

   * Significant valvular or coronary artery disease
   * Uncontrolled hypertension or arrhythmias
   * Primary cardiomyopathies
2. Significant pulmonary disease (FEV1<50% predicted, GOLD III-IV)
3. Inability to exercise or conditions that may interfere with exercise intervention.
4. Myocardial infarction within the last 3 months.
5. Patients with diabetes and/or peripheral vascular disease.
6. Comorbidity that may influence prognosis at one year.
7. Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  he maximum arterial pressure during ventricular systole, measured at the brachial artery by the Mobil-O-Graph using oscillometric technology.
Diastolic Blood Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The minimum arterial pressure during ventricular diastole, measured at the brachial artery by the Mobil-O-Graph using oscillometric technology.
Diastolic Blood Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The average arterial pressure over the cardiac cycle, calculated by the Mobil-O-Graph from oscillometric pressure signals and systolic and diastolic blood pressure values.
Pulse Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The difference between systolic and diastolic brachial blood pressure, calculated by the Mobil-O-Graph and reflecting the pulsatile component of arterial load.
Heart Rate | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The number of heart beats per minute, determined by the Mobil-O-Graph from the time interval between consecutive oscillometric pulse waves.
Central Systolic Blood Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The estimated systolic pressure in the ascending aorta, derived by the Mobil-O-Graph through reconstruction of the central pulse wave from the brachial oscillometric signal.
Central Diastolic Blood Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The estimated diastolic pressure at the central (aortic) level, calculated by the Mobil-O-Graph using pulse wave analysis algorithms.
Central Pulse Pressure | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The difference between estimated central systolic and diastolic blood pressure, calculated by the Mobil-O-Graph to represent aortic pulsatile pressure.
Cardiac Output | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The volume of blood pumped by the heart per minute, estimated by the Mobil-O-Graph from stroke volume calculations combined with heart rate.
Stroke Volume | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The volume of blood ejected by the left ventricle per heartbeat, estimated by the Mobil-O-Graph using hemodynamic modeling based on pulse wave analysis.
Peripheral Vascular Resistance | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  he resistance of the peripheral circulation to blood flow, estimated by the Mobil-O-Graph from calculated mean arterial pressure and cardiac output.
Pulse Wave Velocity | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  The speed at which the arterial pulse wave propagates through the arterial tree, estimated by the Mobil-O-Graph as an indirect marker of arterial stiffness.
Augmentation Index normalized to 75 bpm | Baseline, 0 Minutes post intervention, 30 minutes post intervention, 60 minutes post intervention and 24 hours post intervention
  An index quantifying the contribution of reflected pressure waves to central arterial pressure, estimated by the Mobil-O-Graph from the reconstructed central pulse wave and normalized to a heart rate of 75 beats per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Iván, Cuenca, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: Yes